CLINICAL TRIAL: NCT04568486
Title: Seed-alter Dyad Social Support Intervention for Rural Dwelling Older Adults With T2DM
Brief Title: Social Support Intervention for Older Adults With T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brittany L Smalls (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Brittany L Smalls, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 45777; K01DK116923 (NIH)
Record Dates: First submitted 2020-09-16; First posted 2020-09-29 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rural-dwelling older adults (seed) and Key players (alter (Other): Rural-dwelling older adults will be interviewed to map their social network structure, determine the types of social support provided by members of their social network, and identify key players within these networks. This group will be paired with their key players (identified during interviews) to receive the diabetes education. The pair complete the intervention as a dyad.
  Interventions: Other: Diabetes Empowerment Education Program

INTERVENTIONS:
Other: Diabetes Empowerment Education Program — The Diabetes Empowerment Education Program (DEEP) is an education curriculum designed to help people with pre-diabetes, diabetes, relatives and caregivers gain a better understanding of diabetes self-care. Classes last a total of six weeks, providing participants with eight unique learning modules. Health literacy will be assessed before and after participating in DEEP.

SUMMARY:
This study seeks to describe and evaluate the impact of social support on self-care and clinical outcomes in rural-dwelling older adults with T2DM, test the feasibility and preliminary effectiveness of a 6-week intervention administered by community health workers targeting rural dwelling older adults with T2DM (seed) and an individual within their social support network (alter).

DETAILED DESCRIPTION:
A mixed-methods approach will be used to map social networks of older adults and assess their perceived social support from members of their social network and determine its influence on self-care and clinical outcomes. We will conduct semi-structured interviews with older rural-dwelling adults to map their social network structure, determine the types of social support provided by members of their SN, and identify key players within the older adults' personal network. For this aim, key players are those who can facilitate and promote T2DM self-care on an individual level. These older adults will form a dyad with their alter to participate in a multilevel intervention which includes: gauging the feasibility of using community health workers identified via social network analysis to conduct self-care sessions in rural communities, and the feasibility of seed-alter dyads to provide social support that improves self-care in older adults.

In addition, the seed-alter dyad will participate in 6 weekly sessions of a diabetes education program, led by the community health workers identified previously. Participants will be asked to complete surveys at baseline, 6, and 12 months to assess social support, participants' knowledge about diabetes, and how participants are managing their diabetes.

The preliminary data used for this K01 application was collected from the BRFSS where data is self-reported and its accuracy cannot be confirmed, and a dataset where social support was not the primary objective of the study and there was a small sample size all older adults. Yet, there remains a body of literature that substantiates the influence of social support on T2DM self-care and the disproportionate burden of T2DM in older adults. The proposed research will provide a comprehensive overview of the role of social support and how to leverage this support in a rural community.

ELIGIBILITY:
"Seeds" Inclusion Criteria:

* confirmed diagnosis of T2DM via electronic medical record
* age 65 years or older
* lives within Leslie County
* able to provide consent
* have had at least one clinic visit in the past year

"Seeds" Exclusion Criteria:

* no diagnosis of T2DM via electronic medical record
* under 65 years of age
* unable to speak and understand English
* unable to consent

"Alters" Inclusion Criteria

* 18 years of age or older
* able to provide consent
* has at least weekly contact with the seed

"Alters" Exclusion Criteria

* under 18 years of age
* unable to speak and understand English
* unable to consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Smalls, PhD, Principal Investigator — University of Kentucky
Locations (1):
- UK Center for Excellence in Rural Health, Kentucky Homeplace, Hyden, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seeds: Older adults will be primarily recruited from the University of Kentucky (UK) Center of Excellence in Rural Health clinic.
  Alters: As a result of social network analysis of individual older adults (seeds), a member of the social network (alter) will be identified to participate in as a seed-alter dyad social support intervention.
  The seed and alter must be consented to participate in the intervention.
Period: Overall Study
Arm/Group | Rural-dwelling Older Adults (Seed) and Key Players (Alter
Started | 90
Seed | 65
Alter | 25
Completed | 57
Not Completed | 33
Not completed — Withdrawal by Subject | 26
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Population: Demographics for the seed group were collected for up to 60 participants. Demographics for the alter group were collected for 23 participants
Arm/Group | Rural-dwelling Older Adults (Seed) and Key Players (Alter
Number analyzed (Participants) | 83
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: number of participants with data collected for this demographic
  years
    Seed: number analyzed (Participants) | 60
    Seed | 64.91 (7.66)
    Alter: number analyzed (Participants) | 23
    Alter | 60.52 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: number of participants with data collected for this demographic
  Participants
    seed: number analyzed (Participants) | 57
    seed: Female | 33
    seed: Male | 24
    alter: number analyzed (Participants) | 23
    alter: Female | 16
    alter: Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: data only reported by 3 participants in the seed group and 1 participant in the alter group for this demographic
  Participants
    seed: number analyzed (Participants) | 3
    seed: Hispanic or Latino | 0
    seed: Not Hispanic or Latino | 0
    seed: Unknown or Not Reported | 3
    alter: number analyzed (Participants) | 1
    alter: Hispanic or Latino | 1
    alter: Not Hispanic or Latino | 0
    alter: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: number of participants reporting this demographic
  Participants
    seed: number analyzed (Participants) | 57
    seed: American Indian or Alaska Native | 0
    seed: Asian | 0
    seed: Native Hawaiian or Other Pacific Islander | 0
    seed: Black or African American | 7
    seed: White | 46
    seed: More than one race | 0
    seed: Unknown or Not Reported | 4
    alter: number analyzed (Participants) | 22
    alter: American Indian or Alaska Native | 0
    alter: Asian | 0
    alter: Native Hawaiian or Other Pacific Islander | 0
    alter: Black or African American | 1
    alter: White | 21
    alter: More than one race | 0
    alter: Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 83

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c
Description: The change in participants' hemoglobin A1c measures will be abstracted from their medical records pre- and post-training with the DEEP program. Improved hemoglobin A1c figures suggest an overall success of the DEEP program and a better ability for patients to manage their diabetes.
Time Frame: 12 months
Population: only seed data are reported for this outcome; number of participants measured for this outcome at each time point (56, 21, and 7 respectively)
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | Rural-dwelling Older Adults (Seed) and Key Players (Alter
Number analyzed (Participants) | 60
percentage of hemoglobin
  Baseline: number analyzed (Participants) | 56
  Baseline | 7.004 (1.19)
  6 months: number analyzed (Participants) | 21
  6 months | 6.24 (1.19)
  12 months: number analyzed (Participants) | 7
  12 months | 6.47 (1.05)

2. Secondary Outcome: Systolic Blood Pressure
Description: Participants' systolic and diastolic blood pressures will be abstracted from their medical records pre- and post-training with the DEEP program. Improved blood pressure outcomes suggest an overall success of the DEEP program and a better ability for patients to manage their diabetes.
Time Frame: 12 months
Population: only seed data are reported for this outcome; participants with data for the outcome measure at each time point (58, 21, and 7 respectively)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Rural-dwelling Older Adults (Seed) and Key Players (Alter
Number analyzed (Participants) | 60
mmHg
  Baseline: number analyzed (Participants) | 58
  Baseline | 127.59 (15.23)
  6 months: number analyzed (Participants) | 21
  6 months | 129.57 (17.82)
  12 months: number analyzed (Participants) | 7
  12 months | 129.71 (15.07)

3. Secondary Outcome: Diastolic Blood Pressure
Description: as for outcome 2
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Rural-dwelling Older Adults (Seed) and Key Players (Alter
Number analyzed (Participants) | 60
mmHg
  Baseline: number analyzed (Participants) | 58
  Baseline | 73.59 (11.97)
  6 months: number analyzed (Participants) | 21
  6 months | 77.42 (7.46)
  12 months: number analyzed (Participants) | 7
  12 months | 77.28 (10.59)

4. Secondary Outcome: Lipids
Description: Participants' lipids measures will be abstracted from their medical records pre- and post-training with the DEEP program. Improved lipids outcomes suggest an overall success of the DEEP program and a better ability for patients to manage their diabetes.
Time Frame: 6 weeks
Population: Lipid measures were to be done either using electronic medical records or with a point-of-care (fingerstick) device. Due to HIPAA concerns during IRB approval, investigators decided to rely fully on the fingerstick approach to measuring lipids rather than medical records. At study start up, the fingerstick device intended for use was no longer available for purchase. Therefore, lipids were not collected as part of the study.
Arm/Group | Rural-dwelling Older Adults (Seed) and Key Players (Alter
Number analyzed (Participants) | 0

5. Secondary Outcome: Self-care
Description: The Diabetes self-care management questionnaire consist of 16 questions and sum score was calculated by adding all 16 items. Sum scaled score was computed as actual sum of items/ maximum possible sum of items * 10. The transformed score ranged from 0-10. Higher scores indicating better self-management
Time Frame: 12 months
Population: only seed data are reported for this outcome; participants with data for the outcome measure at each time point (59, 20, and 7 respectively)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rural-dwelling Older Adults (Seed) and Key Players (Alter
Number analyzed (Participants) | 60
score on a scale
  Baseline: number analyzed (Participants) | 59
  Baseline | 6.93 (1.50)
  6 montns: number analyzed (Participants) | 20
  6 montns | 8.08 (1.03)
  12 months: number analyzed (Participants) | 7
  12 months | 8.75 (1.13)

6. Secondary Outcome: Medication Adherence
Description: Participants' medication adherence will be measured from the Brooks Medication Adherence Scale. It measures medication adherence and consists of 6 questions. The total score ranged from 0-6. Less score is associated with being adherent to the medication.
Time Frame: 12 months
Population: only seed data are reported for this outcome; participants with data for the outcome measure at each time point (58, 20, and 7 respectively)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rural-dwelling Older Adults (Seed) and Key Players (Alter
Number analyzed (Participants) | 60
score on a scale
  Baseline: number analyzed (Participants) | 58
  Baseline | 0.84 (1.06)
  6 months: number analyzed (Participants) | 20
  6 months | 0.60 (0.75)
  12 months: number analyzed (Participants) | 7
  12 months | 0.57 (0.78)

7. Secondary Outcome: Health-related Quality of Life Measures
Description: Participants' overall quality of life will be measured with a validated quality of life measure (EuroQol-5D) along 5 dimensions including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The Euro Quality of life questionnaire used 5 questions. The total score was computed by adding the responses for all 5 questions. The total scores ranged from 5 -25. Higher scores is associated with poor quality of life.
Time Frame: 12 months
Population: only seed data are reported for this outcome; participants with data for the outcome measure at each time point (57, 20, and 7 respectively)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rural-dwelling Older Adults (Seed) and Key Players (Alter
Number analyzed (Participants) | 57
score on a scale
  Baseline | 9.45 (3.07)
  6 months: number analyzed (Participants) | 20
  6 months | 9.20 (3.33)
  12 months: number analyzed (Participants) | 7
  12 months | 9.14 (2.67)

ADVERSE EVENTS:
Description: deaths, serious adverse events, and nonserious adverse events were not assessed for study participants
Arm/Group | Rural-dwelling Older Adults (Seed) and Key Players (Alter
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT04568486/Prot_SAP_001.pdf
  • Informed Consent Form (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT04568486/ICF_000.pdf